CLINICAL TRIAL: NCT06835946
Title: Prospective Single-center Observational Trial Aimed at Investigating the Effect of General Anesthesia, Positive Pressure Ventilation and Change of Imaging Modality From Transthoracic Echo to Transesophageal Echo on the Grading of the Severity of Aortic Regurgitation.
Brief Title: Impact of Anesthesia, Positive Pressure Ventilation and Modality of Imaging on the Echocardiographic Assessment of the Severity of Aortic Regurgitation
Status: Recruiting | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Sponsor
Other Study IDs: ANESTIAO
Record Dates: First submitted 2025-02-14; First posted 2025-02-19 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-02

CONDITIONS: Aortic Regurgitation Disease; Aortic Insufficiency
MeSH Terms: conditions — Aortic Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients scheduled for cardiac surgery with previously known aortic regurgitation of any grade

SUMMARY:
The goal of this observational study is to assess the impact of imaging modality (trans-thoracic echo (TTE) vs trans-esophageal echo (TEE)), anesthesia and positive pressure ventilation on the grading of aortic insufficiency.

Patients scheduled for cardiac surgery and in whom a TEE is going to be performed intra-operatively will be enrolled. The grading of the aortic insufficiency will be compared between a TTE performed immediately before the induction of general anesthesia end the TEE performed after induction of general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Known aortic regurgitation of any grade
* Scheduled for a cardiac surgery procedure during which a trans-esophageal echo is planned.

Exclusion Criteria:

* Non sinus rhythm
* Mitral regurgitation more than mild.
* Pre-operative critical state (according to the definition of the EuroSCORE II)
* Presence of a prosthetic aortic valve
* Contra-indication to trans-esophageal echo

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled for cardiac surgery at the "Centre Hospitalier Universitaire de Liège" with any grade of known preoperative aortic regurgitation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Concordance between the grade of aortic regurgitation on pre-operative TTE and intra-operative TEE | From enrollment to the end of the pre-operative trans-esophageal echo
  The preoperative TTE will be performed immediately before anesthesia induction. The intra-operative TEE will be performed after anesthesia induction.
  Five measurements will be used to grade the aortic regurgitation including three major (vena contracta, ration between the width of the aortic regurgitation and the left ventricular outflow tract, and the pressure half time) and two minor (diastolic flow reversal in descending aorta and effective regurgitation orifice area assessed by the proximal isovelocity surface area method).
  The images required to perform these measurements will be acquired three times on non contiguous cardiac cycles at end-expiration. The measurements will be performed offline, by two independent echocardiographers. Each of them will provide a mean for each measurement. The two means will be averaged for each criteria.

SECONDARY OUTCOMES:
Concordance between the grade of aortic regurgitation based on the pre-operative trans-thoracic echo and a trans-thoracic echo repeated immediately after induction of anesthesia. | Enrollment to end of pre-operative trans-thoracic echo
  The aortic regurgitation will be graded similarly as described for the primary outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Liège, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No
The investigators did not consider this when they decided which legal basis would be claimed to collect the data in agreement with the rules of the European general data protection regulation.